CLINICAL TRIAL: NCT00337597
Title: Continuous Regional Analgesia After Total Knee Arthroplasty. Normal Saline or Dextrose 5% in Water as Fluid Medium for Pre-Placement Expansion in Order to Facilitate the Catheter Passing
Brief Title: Continuous Regional Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Charles Pham Dang, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRD 05/7-F
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Analgesia
Keywords: Normal saline; Dextrose 5% in water; neurostimulation; Continuous regional analgesia after total knee arthroplasty
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Other: Glucose 5%
Other: NaCl 0.9%

SUMMARY:
This prospective, comparative and double blind study is aimed to determine if normal saline or dextrose 5% in water will modify the stimulation during the insertion of the stimulating catheter used for continuous femoral and sciatic blocks in total knee replacement.

DETAILED DESCRIPTION:
The operator is blinded to the medium fluid to expand the perineural femoral and sciatic nerves before threading in the stimulating catheter. He records all the electric data of electrolocation of nerve, which will be compared to determine whether or not a difference in intensity is found between normal saline or dextrose 5% in water.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I and II
* Male or non-pregnant female
* 18 - 80 years of age
* Not allergic to iodine or local anesthetics
* Absence of abnormality of coagulation
* Scheduled for total knee replacement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Characteristics of electrolocation of nerve during insertion of the exploring needle and of the stimulating catheter

SECONDARY OUTCOMES:
Efficacy of post-operative analgesia | during 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pham Dang, MD, Principal Investigator — Nantes UH
Locations (2):
- France (2):
  - Departemental Hospital of la Roche sur Yon, La Roche-sur-Yon
  - Nantes University Hospital, Nantes